CLINICAL TRIAL: NCT02780388
Title: A Phase 1b Randomized, Double-blind, Placebo-controlled Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics, and Clinical Response of MEDI4920 in Subjects With Adult-onset Rheumatoid Arthritis
Brief Title: A Phase 1b Study of MEDI4920 in Participants With Adult-onset Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5100C00002; 2015-005318-30 (EudraCT Number)
Record Dates: First submitted 2016-05-03; First posted 2016-05-23 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Adult Onset Rheumatoid Arthritis
Keywords: MEDI4920, VIB4920, CD40L, RA, rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants will receive a single intravascular (IV) dose of placebo matched to VIB4920 (formerly MEDI4920) once every 2 weeks (Q2W) from Day 1 up to 12 weeks.
  Interventions: Other: Placebo
- VIB4920 75 mg (Experimental): Participants will receive a single IV dose of VIB4920 75 mg Q2W from Day 1 up to 12 weeks.
  Interventions: Drug: VIB4920
- VIB4920 500 mg (Experimental): Participants will receive a single IV dose of VIB4920 500 mg Q2W from Day 1 up to 12 weeks.
  Interventions: Drug: VIB4920
- VIB4920 1000 mg (Experimental): Participants will receive a single IV dose of VIB4920 1000 mg Q2W from Day 1 up to 12 weeks.
  Interventions: Drug: VIB4920
- VIB4920 1500 mg (Experimental): Participants will receive a single IV dose of VIB4920 1500 mg Q2W from Day 1 up to 12 weeks.
  Interventions: Drug: VIB4920

INTERVENTIONS:
Drug: VIB4920 — Participants will receive a single IV dose of VIB4920 Q2W from Day 1 up to 12 weeks.
  Other Names: MEDI4920
  Arms: VIB4920 1000 mg; VIB4920 1500 mg; VIB4920 500 mg; VIB4920 75 mg
Other: Placebo — Participants will receive a single IV dose of placebo matched to VIB4920 Q2W from Day 1 up to 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether VIB4920 (formerly MEDI4920) is safe and well tolerated in participants with adult-onset rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024. Originally Viela Bio was the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* adult-onset rheumatoid arthritis
* swollen and tender joints

Exclusion Criteria:

* venous thromboembolism or arterial thrombosis
* pregnant or breastfeeding
* positive hepatitis B, hepatitis C, and human immunodeficiency virus infection
* active or untreated latent tuberculosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (8):
  - Research Site, Anniston, Alabama
  - Research Site, DeBary, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, South Miami, Florida
  - Research Site, Cincinnati, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Mesquite, Texas
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Poznan
  - Research Site, Warsaw

REFERENCES:
- [Result] Karnell JL, Albulescu M, Drabic S, Wang L, Moate R, Baca M, Oganesyan V, Gunsior M, Thisted T, Yan L, Li J, Xiong X, Eck SC, de Los Reyes M, Yusuf I, Streicher K, Muller-Ladner U, Howe D, Ettinger R, Herbst R, Drappa J. A CD40L-targeting protein reduces autoantibodies and improves disease activity in patients with autoimmunity. Sci Transl Med. 2019 Apr 24;11(489):eaar6584. doi: 10.1126/scitranslmed.aar6584. PMID 31019027
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/31019027?report=abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 12 May 2016 to 09 Aug 2018 in Poland and the United States of America.
Pre-assignment Details: A total of 117 participants were screened in the study, out of which 60 were screen failures. A total of 57 participants were randomized in this study.
Groups:
- Placebo: Participants received a single intravascular (IV) dose of placebo matched to VIB4920 (formerly MEDI4920) once every 2 weeks (Q2W) from Day 1 up to 12 weeks.
- VIB4920 75 mg: Participants received a single IV dose of VIB4920 75 mg Q2W from Day 1 up to 12 weeks.
- VIB4920 500 mg: Participants received a single IV dose of VIB4920 500 mg Q2W from Day 1 up to 12 weeks.
- VIB4920 1000 mg: Participants received a single IV dose of VIB4920 1000 mg Q2W from Day 1 up to 12 weeks.
- VIB4920 1500 mg: Participants received a single IV dose of VIB4920 1500 mg Q2W from Day 1 up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Started | 15 | 8 | 10 | 12 | 12
Completed | 14 | 6 | 10 | 12 | 12
Not Completed | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to treat population included all randomized and treated participants, grouped according to assigned treatment.
Groups:
- Placebo: Participants received a single intravascular (IV) dose of placebo matched to VIB4920 once every 2 weeks (Q2W) from Day 1 up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg | Total
Number analyzed (Participants) | 15 | 8 | 10 | 12 | 12 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.0) | 57.9 (7.4) | 53.7 (9.8) | 52.1 (11.5) | 50.9 (8.6) | 54.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 6 | 10 | 10 | 46
  Male | 1 | 2 | 4 | 2 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 1 | 0 | 7
  Not Hispanic or Latino | 12 | 6 | 9 | 11 | 12 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 2 | 0 | 5
  White | 13 | 8 | 9 | 10 | 12 | 52
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 169
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 15 | 8 | 10 | 12 | 12
Participants
  TEAEs | 13 | 3 | 7 | 6 | 10
  TESAEs | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent AEs of Special Interests (AESIs)
Description: An AESI (serious or non-serious) is one of scientific and medical interest specific to understanding of study drug and may have required close monitoring, collection of additional information by investigator and rapid communication by investigator to the sponsor.
Time Frame: Day 1 through Day 169
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 15 | 8 | 10 | 12 | 12
Participants
  Encephalitis | 0 | 0 | 0 | 0 | 1
  Herpes simplex | 0 | 0 | 0 | 0 | 1
  Oral herpes | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of VIB4920
Description: Maximum observed plasma concentration (Cmax) of VIB4920 is reported.
Time Frame: Dose 1: Post-dose (end of infusion) on Day 1, pre-dose on Day 15; Dose 7: Pre- and post-dose (end of infusion) on Day 85; and on Days 92, 99, 113, 141, and 169
Population: Pharmacokinetics (PK) population included all treated participants with at least one PK sample with detectable VIB4920. Participants with available PK sample at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
µg/mL
  Dose 1 | 20.6 (5.26) | 158 (95.4) | 392 (84.4) | 360 (83.8)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 24.4 (3.72) | 157 (40.7) | 423 (114) | 627 (159)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of VIB4920
Description: Time to maximum plasma concentration (Tmax) of VIB4920 is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
Days
  Dose 1 | 0.02 [0.02 to 1.00] | 0.04 [0.04 to 0.04] | 0.06 [0.06 to 1.00] | 0.06 [0.06 to 0.06]
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 0.02 [0.02 to 0.02] | 0.04 [0.04 to 0.04] | 0.06 [0.06 to 0.06] | 0.06 [0.06 to 0.06]

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve of the Dosing Interval (AUCtau) of VIB4920
Description: Area under the plasma concentration time curve of the dosing interval (AUCtau) of VIB4920 is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
µg*day/mL
  Dose 1 | 122 (25.5) | 669 (164) | 2150 (496) | 2360 (466)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 262 (94.7) | 1430 (466) | 3760 (1370) | 5850 (1530)

6. Secondary Outcome: Dose Normalized AUCtau of VIB4920
Description: Dose normalized AUCtau of VIB4920 is reported. Dose normalized AUCtau is calculated by dividing AUCtau by the dose of administered VIB4920 (in mg).
Time Frame: as for outcome 3
Population: Pharmacokinetics (PK) population included all treated participants with at least one PK sample with detectable VIB4920. Participants with available PK sample at specified time points were analysed.
Measure: Mean (Standard Deviation); unit: µg*day/mL/mg
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
µg*day/mL/mg
  Dose 1 | 1.62 (0.341) | 1.34 (0.328) | 2.15 (0.496) | 1.58 (0.311)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 3.49 (1.26) | 2.87 (0.931) | 3.76 (1.37) | 3.90 (1.02)

7. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of VIB4920
Description: Area under the plasma concentration time curve from time zero to extrapolated infinite time (AUC0-inf) of VIB4920 is reported.
Time Frame: Post-dose (end of infusion) on Day 1, pre-dose on Day 15; pre- and post-dose (end of infusion) on Day 85; and on Days 92, 99, 113, 141, and 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 7 | 10 | 10 | 12
µg*day/mL | 163 (42.7) | 824 (228) | 2660 (744) | 3480 (842)

8. Secondary Outcome: Systemic Clearance (CL) of VIB4920
Description: Systemic clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
mL/day
  Dose 1: number analyzed (Participants) | 7 | 10 | 10 | 12
  Dose 1 | 489 (135) | 654 (203) | 405 (120) | 457 (120)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 449 (129) | 536 (152) | 421 (107) | 381 (94.8)

9. Secondary Outcome: Terminal Elimination Half-life (t½) of VIB4920
Description: Terminal elimination half-life (t½) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
Days
  Dose 1: number analyzed (Participants) | 7 | 10 | 10 | 12
  Dose 1 | 6.25 (1.26) | 5.61 (0.891) | 6.12 (0.725) | 8.70 (2.61)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 7.82 (1.50) | 9.58 (1.57) | 9.72 (1.32) | 9.58 (1.37)

10. Secondary Outcome: Volume of Distribution at Steady State (Vss) of VIB4920
Description: Volume of distribution at steady state (Vss) of VIB4920 is reported.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 8 | 10 | 12 | 12
mL
  Dose 1 | 4230 (595) | 5040 (1220) | 3510 (844) | 5380 (1210)
  Dose 7: number analyzed (Participants) | 6 | 10 | 12 | 11
  Dose 7 | 5060 (980) | 5600 (1010) | 4620 (1060) | 4100 (905)

11. Secondary Outcome: Accumulation Ratio (AR) of VIB4920
Description: Accumulation ratio of VIB4920 is reported. Accumulation ratio was determined using AUCtau, Dose 7/AUCtau, Dose 1.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 6 | 10 | 12 | 11
Ratio | 1.51 (0.265) | 1.51 (0.287) | 1.20 (0.251) | 1.76 (0.305)

12. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) Titer to VIB4920
Description: The number of participants with positive antibodies to VIB4920 are reported.
Time Frame: Pre-dose on Days 1, 29, 57, and 85; and on Days 141, and 169
Population: Intent-to treat population included all randomized and treated participants, grouped according to assigned treatment. Participants with available ADA sample were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
Number analyzed (Participants) | 6 | 10 | 12 | 12
Participants | 3 | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 169
Arm/Group | Placebo | VIB4920 75 mg | VIB4920 500 mg | VIB4920 1000 mg | VIB4920 1500 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8 | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8 | 0/10 | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 13/15 | 3/8 | 7/10 | 6/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | VIB4920 75 mg (N=8) | VIB4920 500 mg (N=10) | VIB4920 1000 mg (N=12) | VIB4920 1500 mg (N=12)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | VIB4920 75 mg (N=8) | VIB4920 500 mg (N=10) | VIB4920 1000 mg (N=12) | VIB4920 1500 mg (N=12)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral small vessel ischemic disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Viela Bio has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multicentre publication.

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02780388/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT02780388/SAP_001.pdf